CLINICAL TRIAL: NCT03665233
Title: Virtual Reality for Post Operative Pain Management After Total Knee Arthroplasty: a Randomized, Controlled, Multi-center, Double Blind, Parallel Group, Superiority Trail to Evaluate VR as a Component of a Multi-modal Pain Treatment
Brief Title: Virtual Reality for Post Operative Pain Management After Total Knee Arthroplasty
Acronym: VR4POPKA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients (covcid restrictions)
Sponsor: Clinique Saint-Jean, Bruxelles (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Dr. Arnaud Bosteels, Head of the anaesthesia department, principal investigator, Clinique Saint-Jean, Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VRAB001; 2018-001559-10 (EudraCT Number)
Record Dates: First submitted 2018-09-02; First posted 2018-09-11 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Virtual Reality; Pain, Postoperative; Knee Arthropathy; Anesthesia; Hypnosis
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sh-group (Sham Comparator): The patients in this arm get standard treatment, together with a sham version of a VR session.
  Interventions: Device: VR
- VR-group (Active Comparator): These patients get a VR session with the standard treatment
  Interventions: Device: VR

INTERVENTIONS:
Device: VR — People in the VR-group get a VRH session during the CPM physiotherapy , people in the sham group get a VR sham session, while they both can enjoy Standard Treatment
  Other Names: Aqua VRH session; Oncomfort; Gear VR

SUMMARY:
Virtual reality has been used for acute pain management (burn patients) with positive results. Hypnosis has known beneficial effects on patients in the peri-operative setting. The investigators are combining both by giving a virtual reality hypnosis (VRH) session to the patients during a known painful post-operative moment. (physiotherapy) It is the investigator intention to compare pain after physiotherapy during the first 3 days after a total knee arthroplasty, between 2 groups. One group , the VR group gets standard treatment with VRH and the second, the sham group, gets standard treatment with a sham VR session.

DETAILED DESCRIPTION:
Introduction: Postoperative pain frequently occurs after total knee arthroplasty. The IASP defines pain as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage". Pain is a major cause of post-operative distress and has a variety of side effects and complications. Chronic post surgical pain is probably the most feared complication of acute pain. Therefore, adequate pain control after surgery is mandatory.

In modern western healthcare, multi-modal pain treatment is the standard of care. This means that a variety of drugs, acting on different receptors, are used alongside non-pharmacological interventions, to decrease pain. Such an approach enables the physician to use a lower concentration of a specific drug, in order to avoid adverse effects that can occur when giving higher doses of one individual drug. These drugs are based on the analgesic ladder of the WHO to relief cancer pain. From the different drugs that are used, the major concern will be with the opioids, as they are known to have major complications. Especially today in the USA there is an epidemic of opioid related deaths. Very often these drugs have been prescribed in a post-operative setting. The search for a different non-pharmacological analgesic treatment is today, more than ever, a pressing need.

Virtual reality (VR) is a non-pharmacological way to decrease pain in a number of different situations. It has been around for some years, some articles describing VR in medicine are 25 years old but it only recently became a popular medical treatment since the introduction of the Oculus Rift in 2014. Before that HMDs (head-mounted display) were expensive and very bulky devices. Since the introduction of the Oculus Rift HMD the availability and usability of VR has increased dramatically.

In the post-operative period pain at rest is generally reported to be acceptable by our patients (VAS<3), but if movements are involved the pain increases to unacceptable levels. Postoperative physiotherapy generally involves the use of a continuous passive motion (CPM), a machine used for passive bending of the knee. This postoperative mobilization is one of the major causes of pain in the aftermath of a total knee arthroplasty.

Available evidence: Virtual Reality (VR) has been shown to reduce pain in different situations. From experimental pain in healthy subjects to changing dressing of burn patients, several studies have shown the use of immersive VR therapy as an adjunct for pain treatment.

The use of VR in children has frequently been studied, as it decreases pain and anxiety during painful medical procedures.

The combination of VR and standard treatment (ST) has shown to have a superior analgesic efficacy compared to VR or ST alone .

In the medical VR world there are different types of applications. Some of these act as "distractors" (playing games, looking at natural scenery) and some have included elements of therapeutic hypnosis. With these applications the patients are (self)-induced in a hypnotic state.

Medical hypnosis has been shown to have a tremendous impact on post-operative recovery, reducing anxiety and pain. Medical hypnosis is a one on one intervention, making it time and labor consuming and people using hypnosis need to be well trained to perform the technique safely. Bringing a patient in a hypnotic state can only be achieved by using appropriate verbal quotes and this can be problematic if the patient speaks another language.

Although the surgical population would benefit greatly by using medical hypnosis, only few patients are offered this technique.

Using a VR application with therapeutic hypnotic elements can be a great way to share with many patients the positive effects of hypnotic therapy.

Trial : the investigators decided therefore to use a medical VR application that includes therapeutic hypnotic elements. They want to compare the analgesic efficacy of standard treatment with medical virtual reality and standard treatment with a sham VR session in postoperative pain management, after the patient have had a session of physiotherapy, as this is a painful moment in the post operative period. Using a sham VR session is lickely to produce some sort of analgesia as any disctraction with VR can have a positive effect. But this sham session isn't an enjoyable VRH session, therefore the authors still expect a significant difference in pain reduction.

Using the sham seems inevitbale because it is not possible to blind the patients otherwise to their own traetment. If the authors would use use a control group there would be a high risk of biais because of the dissapointement for the patients not receiving any VR.

Each includable patient will be approached before the day of surgery and asked for participation in the study, after verifying the absence of any exclusion criteria.

The investigators will present the study to the patients, using a patient oriented explicatory form, after which they will look at the informed consent together with the patient. If necessary they will give the patient some time to reflect and come back after a while, to sign and collect, or not, the informed consent.

Randomization will be done earlier using a web based block randomization program : www.randomization.com Each patient will be assigned to either a standard treatment with VR sham group (Sh-group) or a standard treatment with Virtual reality group (VR-group). The virtual reality will be an application designed by Oncomfort®. It is a session called AQUA, which includes an underwater experience guided by a whale. The VR sham experience is also an underwater based experience but without any coherence between the different images. The HMD is a VR Gear from Samsung-Oculus and the mobile phone used is a Samsung Galaxy 7.

Interventions happen on the day of surgery (DOS), on post operative day 1-2 and 3 (POD1, POD2 and POD3. )

On the day of surgery :

Before going to the OR each included patient (both VR and Sh group) fills in a STAI Y questionnaire gives a VAS pain score Before going to the OR, patients in the VR group get additionally a 45 min session of VR : AQUA and patients in the Sh group get 45 min of a sham session.

Each patient gets a TKA. There is no interference with the anaesthesia protocol. This is, as usual, decided between the patient and the anaesthetist working in the OR. Some parts of the peri-operative and the post-operative protocols however are standardized:

Peroperative General anesthesia Paracetamol 1g every 6 h If there are no contra-indications : anti-inflammatory drugs (ketorolac) 3x/d IV, (including a PPI (proton pump inhibitor) if necessary) Dexamethasone 0,5 -1 mg/kg Tranexamic acid 1 g Use of a tourniquet by the surgeon Infiltration of the posterior part of the knee by the surgeon with levobupivacaine 0.2% PCIA Morphine Femoral nerve block single shot (with 15 ml levobupivacaine 0,25% ) , before the start of the surgery Postoperative Paracetamol Anti-inflammatory drugs PCIA morphine Ice application 3 times a day Rescue medication : Tramadol 50 mg, max 6 per day

POD1-POD2 -POD3 During the post operative days patients get passive mobilization of the knee with the CPM device (Kinetec).

During this exercise patients in the VR-group get a 45 minute VR session and teh Sh-group gets a 45 min sham session. The physiotherapist (who gets a specific training) or another investigator will put on the mask. The CPM device starts 10 min after the start of the VR session. All the patients get standard care, which means they can use their PCIA morphine, as required.

After each session a blinded investigator measures the VAS pain score, the anxiety score with the STAY-I questionnaire and the morphine consumed.

On POD3 or on the day of discharge (if earlier) patients will be asked to rate their satisfaction (with a VAS). The physiotherapist will also rate their appreciation of the functional rehabilitation, by comparing the increase of passive flexion between POD1 and POD3.

Total morphine consumption (until POD3) and length of stay will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a TKA
* General anesthesia and single shot fem block
* Adults (> 18 years)
* Elective procedures

Exclusion Criteria:

* Refusal of consent
* History of seizures
* History of drug abuse
* History of psychiatric diseases
* Patients with impaired hearing
* Patients with impaired vision
* Patients afraid of submarine worlds
* Chronic pain patients
* Claustrophobia
* Language not available on VR system

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
The comparison of opioid consumption after physiotherapy, when using VRH or VR sham | on post operative day 1
  After each physiotherapy session with continuous passive movement (CPM), a blinded investigator will measure the opioid consumption .
The comparison of opioid consumption after physiotherapy, when using VRH or VR sham | on post operative day 2
  After each physiotherapy session with continuous passive movement (CPM), a blinded investigator will measure the opioid consumption
The comparison of opioid consumption after physiotherapy, when using VRH or VR sham | on post operative day 3
  After each physiotherapy session with continuous passive movement (CPM), a blinded investigator will measure the opioid consumption

SECONDARY OUTCOMES:
The change in anxiety measured with an anxiety scale, after physiotherapy, between the control (standard treatment ) and the VR group (standard + VR treatment) | on post operative day (POD) 1-2-3
  After each physiotherapy session with CPM, a blinded investigator will measure the anxiety using STAI Y. The State Trait Anxiety Inventory. This is a questionnaire of 20 questions assessing a patients state of anxiety. The answer to every questions can be rated from 1 until 4. The high rthe score the higher the anxiety.
The variation in patient satisfaction at the end of the third day, between the participants using the VRH or not. | on post operative day (POD) 3
  after post operative day 3 a blinded investigator will measure the satisfaction score using (VAS) visual analogue scale. This is a scale going from no satisfaction at all until the best satisfaction one can imagine. The scale is like a horizontal yardstick with a cursor and the patient is asked to move to cursor to the level of his satisfaction. On the other side of the scale is a metric system from 0-10 cm. This way the satisfaction can be scored out of 10. The higher the number the better the satisfaction.
The comparison in pain after post-operative physiotherapy using VAS | on post operative day 1-2-3
  a blinded investigator will measure the VAS pain score after each physiotherapy session involving a CPM.This is a scale going from no satisfaction at all until the best satisfaction one can imagine. The scale is like a horizontal yardstick with a cursor and the patient is asked to move to cursor to the level of his satisfaction. On the other side of the scale is a metric system from 0-10 cm. This way the pain can be scored out of 10. The higher the number the worser the pain
The comparison of the evolution of the knee flexion with the CPM (Continuous passive motion) when using VRH or not | on post operative day 1 and 3
  Measure the increase of flexion of the knee on the CPM device between POD1 and POD3
The variance in the length of stay after a total knee arthroplasty between the treatment and the control group. | This will be assessed 1 week after surgery
  measuring the length of stay at the hospital, from the day (and hour) of surgery, until the patient is ready for discharge (day and hour). This is the moment the operator decides that the patient is fit enough to leave the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bosteels, MD, Principal Investigator — Clinique Saint Jean Brussels
Locations (1):
- Clinique Saint Jean, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No